CLINICAL TRIAL: NCT03802903
Title: Efficacy and Safety of Remo-Wax for Removal of Impacted Earwax; an Open, Single-arm, Non-randomised, Multicentre Clinical Study
Brief Title: Efficacy and Safety of Remo-Wax for Removal of Impacted Earwax
Acronym: Remo-Wax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3126001
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Cerumen Impaction of Both Ears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remo-Wax (Experimental): Test product will be applied into ear canal for 20-60 minutes.
  Interventions: Device: Remo-Wax

INTERVENTIONS:
Device: Remo-Wax — topical treatment

SUMMARY:
The study evaluates if Remo-Wax ear drops can soften impacted earwax.

DETAILED DESCRIPTION:
This is an open, single-arm multicentre study to confirm the efficacy and safety of a commercially available Remo-Wax ear drops containing allantoin for dissolving and removing impacted earwax. Subjects that qualify for enrollment and provide informed consent wil be treated with topical earwax softening product.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Male or female patients over 1 year old who have cerumen impaction.
3. Presence of excessive or impacted cerumen [excessive or impacted cerumen is identified as causing partial (> 50%) or complete occlusion of at least one ear canal when attempting to visualize the tympanic membrane.

Exclusion Criteria:

1. Hypersensitivity to any product ingredient(s) or history of anaphylactic/anaphylactoid reactions.
2. History of tympanic membrane perforation, tympanostomy tubes, or otitis externa in the previous 6 months.
3. External ear infection.
4. Middle ear infection
5. Past ear surgery.
6. Otorrhea.
7. Temporal bone neoplasm.
8. Presence of known or suspected mastoiditis.
9. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data (e.g. ear eczema or seborrhoea, ear canal stenosis, exostoses).
10. Deafness in the contralateral ear (single sided deafness).
11. Use of any ototopical drug or cerumen-removal product (with the exception of water or physiologic saline) during the preceding 3 days.
12. Use of hearing aids.
13. Participation in another drug study within 60 days prior to the start of the present study.
14. Predictable poor compliance or inability to communicate well with the investigator.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Tympanic membrane visuality | 20-60 minutes
  Tympanic membrane will be assessed in five grades of occlusion's severity after each treatment application.
  Normal - insignificant earwax present, Minimal - minimal impacted cerumen in ear canal, Mild - some impacted cerumen in ear canal, Moderate - moderate impacted cerumen in ear canal, Severe - excessive impacted cerumen in ear canal

CONTACTS AND LOCATIONS:
Locations (1):
- LOR Clinic, Vilnius, Lithuania